CLINICAL TRIAL: NCT02388997
Title: An Evaluation of Treatment With Omalizumab to Improve the Asthmatic Response to an Experimental Infection With Rhinovirus
Brief Title: Treatment With Omalizumab to Improve the Asthmatic Response to Rhinovirus Experimental Infection With Rhinovirus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Peter Heymann, MD, Head, Pediatric Allergy/Immunology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14427; U01AI100799 (NIH)
Record Dates: First submitted 2015-03-09; First posted 2015-03-17 (Estimated); Results first posted 2018-07-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Asthma
Keywords: mild asthma; young adults; rhinovirus
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mild asthmatics treated with omalizumab (Active Comparator): Subjects with mild asthma will be treated with omalizumab for 8 weeks before and for 3 weeks after an experimental challenge with rhinovirus. Omalizumab will be given subcutaneously every 2 to 4 weeks according to the manufacturer's recommendations.
  Interventions: Drug: omalizumab; Biological: Rhinovirus (strain 16)
- Mild asthmatics treated with placebo medication (Placebo Comparator): Subjects with mild asthma will be treated with placebo medication for 8 weeks before and for 3 weeks after an experimental challenge with rhinovirus. The placebo mediation will consist of the same diluent used for suspending the omalizumab without omalizumab added.
  Interventions: Drug: omalizumab; Biological: Rhinovirus (strain 16)

INTERVENTIONS:
Drug: omalizumab — This medication has been approved for clinical use to treat patients with moderate to severe asthma by the FDA in 2003 and for use in this study (BB-IND# 10510)
  Other Names: Xolair
Biological: Rhinovirus (strain 16) — This strain of pooled rhinovirus has been approved for use in experimental challenges (BB-IND# 15162) and for use in this study (BB-IND# 10510) by the FDA.

SUMMARY:
Population surveys have shown a positive correlation between increased levels of total serum immunoglobulin E (IgE) and bronchial hyperreactivity. However, it is also clear that exacerbations of asthma are frequently triggered by viral respiratory tract infections, especially those caused by human rhinovirus (RV), also known as the "common cold" virus. This protocol explores the relationship between rhinovirus and allergen/IgE provoked inflammation. Experimental challenges with human (RV) result in more persistent upper respiratory tract symptom scores in asthmatics than in controls. Asthmatics with high levels of IgE also show greater sensitivity to methacholine and higher levels of expired nitric oxide (eNO) than those with low levels of IgE. These data suggest that patients with asthma and high levels of IgE are more likely to have pre-existing inflammation of the airways before virus challenge. This study is being done to determine whether anti-IgE therapy (with omalizumab) will lead to a significant decline in inflammatory biomarkers prior to virus inoculation, and thus reduce the severity of clinical manifestations after an experimental human RV challenge.

DETAILED DESCRIPTION:
The study is a randomized, double-blind placebo controlled study involving a group of 42 mild asthmatics. Subjects will be randomized 1:1 to omalizumab (a humanized monoclonal anti-IgE antibody) or placebo for 8 weeks and then inoculated with rhinovirus (strain-16 produced under GMP conditions and approved for this research by the FDA). Clinical and laboratory (mechanistic) data will be evaluated for 8 weeks before and for 4 weeks after the virus challenge.

The study is being done to test the hypothesis that the reduction of total free IgE in asthmatics treated with omalizumab for 8 weeks prior to and during an experimental RV challenge will lead to a significant decline in lower respiratory tract (chest) symptoms recorded by subjects during the first four days of infection following the challenge compared to lower respiratory tract symptoms recorded during the same period by asthmatic subjects who are treated with placebo.

The primary endpoint will be based on the comparison of cumulative lower respiratory tract symptoms scores (CLRTS) in the asthmatic subjects treated with omalizumab compared to those treated with placebo over the first 4 days of acute infection. Diary cards will be scored daily for cough, shortness of breath, chest discomfort and wheezing using a modification of the Jackson criteria. To participate in this study, subjects must live within 90 minutes by car from the University of Virginia.

Note: This protocol has been reviewed and is being monitored for safety by the NIH/NIAID Safety Monitoring Committee and by he IRB at the University of Virginia (IRB-HSR# 14427).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to understand and provide written informed consent
* Age 18 to 40 years of age, any gender, any racial/ethnic origin
* Physician-diagnosed asthma
* Asthma Control Test (ACT) score > 19
* Short-acting beta-agonist use < daily in last 4 weeks
* Forced expired volume at 1 second (FEV1) > 70%, or FEV1/FVC ratio > 75% for subjects with forced vital capacity (FVC) values between 80 and 87% predicted whose FEV1 values fall below 70%.
* Positive Methacholine challenge test (i.e. at least 20% fall in FEV1 at a Methacholine concentration of ≤16 mg/ml) at screening protocol before enrollment.
* Total serum IgE level greater than or equal to 125 IU/ml evaluated during screening protocol.
* Positive test for allergic sensitization by prick skin testing documented during screening protocol. to allergens associated with current allergen exposure at the time of the rhinovirus (RV) challenge: e.g., dust mite, Alternaria, and/or ragweed for subjects challenged with RV in the fall, or positive tests to tree and/or grass pollen allergens for those challenged with RV in the spring. In keeping with the study design goals of inoculating subjects during periods of allergen exposure, sensitization to other allergens (e.g., cat or dog) will also qualify for enrollment if subjects are currently exposed to these allergens at home.

Participant must be willing to comply with study procedures and requirements.

-

Exclusion Criteria:

* Inability or unwillingness of a participant or subject's legal representative to give written informed consent and HIPPA authorization
* Positive test for serum neutralizing antibody to rhinovirus (strain-16) at screening within 6 weeks (i.e., subjects with a neutralizing antibody titer > 1:4 will be excluded).
* To avoid RV-16 inoculations in subjects with more restrictive lung volumes, those whose FVC is < 80% predicted will also be excluded.
* Total IgE levels measured at screening protocol that are too elevated based on a subjects weight, to meet the recommendations for treatment with Omalizumab.
* Chronic heart disease, lung diseases other than asthma, or other chronic illnesses, including primary and/or secondary immunodeficiency.

Hospitalization or treatment in the ER for asthma (unless the treatment involved the use of a bronchodilator only) during the last three years.

* Subjects who have had one or more night time awakenings caused by asthma symptoms and/or who have needed their short acting beta-2 agonist (SABA; e.g., albuterol) inhaler for asthma symptoms > 4 days during the week before enrollment, or during the week before the virus challenge.
* Intubation or management in the intensive care unit for an asthma exacerbation
* An upper or lower respiratory tract infection within six weeks prior to enrollment
* Previous nasal or sinus surgery within the last 12 months.
* Who have a 5 pack/year history of smoking, or any smoking within the last 6 months.
* Female subjects who are, or who plan to become, pregnant during the study, or who are nursing a baby. Additionally, to be included in this study, a woman of child-bearing potential must have a negative urine pregnancy test at screening, during the run, and prior to viral inoculation and agree to use an effective method of birth control such as, but not limited to, birth control pills, contraceptive foam, diaphragm, intra uterine device (IUD), abstinence, or condoms.
* Subjects who have used omalizumab within 12 months prior to enrollment, or inhaled corticosteroids,inhaled ipratropium bromide, an inhaled long acting beta agonist, inhaled cromolyn or nedocromil or systemic leukotriene modifiers for their asthma on a daily basis within 4 weeks prior to enrollment or subjects using nasal corticosteroids on a daily basis within 4 weeks prior to enrollment. Subjects who are currently receiving beta-adrenergic blocking agents.
* Subjects who are currently receiving allergen immunotherapy (IT), or who have received allergen IT within the last 3 years.
* Hemoglobin <11.5 g/dL for non-African American subjects or hemoglobin < 11.0 g/dL for African American subjects detected during screening within 6 weeks of enrollment.
* Absolute neutrophil count (ANC) < 1800 cells/mm3 (or 1.8 K/uL) detected during screening within 6 weeks of enrollment or prior to virus inoculation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter W Heymann, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mild Asthmatics Treated With Omalizumab | Mild Asthmatics Treated With Placebo Medication
Started | 15 | 16
Completed | 12 | 10
Not Completed | 3 | 6
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lung function exclusion criteria | 0 | 2
Not completed — Tested positive for virus during run-in | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild Asthmatics Treated With Omalizumab | Mild Asthmatics Treated With Placebo Medication | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Full Range); unit: years] | 20.4 [18 to 28] | 22.8 [18 to 33] | 21.6 [18 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 6 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 2 | 3
  White | 11 | 12 | 23
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Total serum IgE level (IU/ml) [Geometric Mean (Full Range); unit: IU/ml] | 238 [133 to 493] | 266 [140 to 529] | 252 [133 to 529]
Negative serum neutralizing antibody to rhinovirus-16 [Count of Participants; unit: Participants] | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Airway Symptom Scores Experienced by Participants During the First 4 Days of the Acute Infection.
Description: The primary outcome was based on the comparison of cumulative lower respiratory tract symptoms scores (CLRTS) in the asthmatic subjects treated with omalizumab compared to those treated with placebo over the first 4 days of acute infection. The symptoms evaluated daily included wheeze, chest tightness, and shortness of breath. Symptom scores were recorded by subjects twice daily (in the morning and evening). Each symptom was scored on a scale of 1 to 3. Therefore, the total maximum (worst) score for a day would be 18. The scores recorded daily could range from 0 to 18.
Time Frame: 4 days
Population: Two participants in the mild asthmatics treated with omalizumab treatment arm had to be dropped according to protocol because one developed a positive qPCR test for rhinovirus (the virus used for inoculation) 4 weeks before virus inoculation, and the other developed a positive qPCR test for rhinovirus during the week before inoculation.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mild Asthmatics Treated With Omalizumab | Mild Asthmatics Treated With Placebo Medication
Number analyzed (Participants) | 10 | 10
units on a scale | 4.0 [0 to 5.0] | 3.3 [0 to 7.4]
Statistical Analysis 1: Comparison: Mild Asthmatics Treated With Omalizumab vs Mild Asthmatics Treated With Placebo Medication; Test type: Superiority; p = 0.59, 2-sample t-test with unequal variences

2. Secondary Outcome: Airway Symptom Scores Experienced by Participants During the First 7 Days of the Acute Infection.
Description: This secondary outcome was based on the comparison of cumulative lower respiratory tract symptoms scores (CLRTS) in the asthmatic subjects treated with omalizumab compared to those treated with placebo over the first 7 days of acute infection. The symptoms evaluated daily included wheeze, chest tightness, and shortness of breath. Symptom scores were recorded by subjects twice daily (in the morning and evening). Each symptom was scored on a scale of 1 to 3. Therefore, the total maximum (worst) score for a day would be 18. The scores recorded daily could range from 0 to 18.
Time Frame: 7 days
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mild Asthmatics Treated With Omalizumab | Mild Asthmatics Treated With Placebo Medication
Number analyzed (Participants) | 10 | 10
units on a scale | 5.0 [0 to 12.8] | 8.4 [0 to 18.4]
Statistical Analysis 1: Comparison: Mild Asthmatics Treated With Omalizumab vs Mild Asthmatics Treated With Placebo Medication; Test type: Superiority; p = 0.58, 2-sample t-test with unequal variances

3. Secondary Outcome: Airway Symptom Scores Experienced by Participants During the 21 Days of Monitoring During the Infection.
Description: This secondary outcome was based on the comparison of cumulative lower respiratory tract symptoms scores (CLRTS) in the asthmatic subjects treated with omalizumab compared to those treated with placebo over the 21 days of monitoring during the infection. The symptoms evaluated daily included wheeze, chest tightness, and shortness of breath. Symptom scores were recorded by subjects twice daily (in the morning and evening). Each symptom was scored on a scale of 1 to 3. Therefore, the total maximum (worst) score for a day would be 18. The scores recorded daily could range from 0 to 18.
Time Frame: 21 days
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mild Asthmatics Treated With Omalizumab | Mild Asthmatics Treated With Placebo Medication
Number analyzed (Participants) | 10 | 10
units on a scale | 19.9 [0 to 49.7] | 17.0 [0 to 41.0]
Statistical Analysis 1: Comparison: Mild Asthmatics Treated With Omalizumab vs Mild Asthmatics Treated With Placebo Medication; Test type: Superiority; p = 0.87, 2-sample t-test with unequal variances

4. Secondary Outcome: Airway Symptom Scores Experienced by Participants During the First 4 Days of the Acute Infection With Cough.
Description: This secondary outcome was based on the comparison of cumulative lower respiratory tract symptoms scores (CLRTS) in the asthmatic subjects treated with omalizumab compared to those treated with placebo over the first 4 days of acute infection. The symptoms evaluated daily included wheeze, chest tightness, shortness of breath and cough. Symptom scores were recorded by subjects twice daily (in the morning and evening). Each symptom was scored on a scale of 1 to 3. Therefore, the total maximum (worst) score for a day would be 24. The scores recorded daily could range from 0 to 24.
Time Frame: 4 days
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mild Asthmatics Treated With Omalizumab | Mild Asthmatics Treated With Placebo Medication
Number analyzed (Participants) | 10 | 10
units on a scale | 3.7 [0 to 7.5] | 5.3 [0.7 to 9.9]
Statistical Analysis 1: Comparison: Mild Asthmatics Treated With Omalizumab vs Mild Asthmatics Treated With Placebo Medication; Test type: Superiority; p = 0.55, 2-sample t-test with unequal variances

5. Secondary Outcome: Airway Symptom Scores Experienced by Participants During the First 4 Days of the Acute Infection (Upper Respiratory Tract Symptoms).
Description: This secondary outcome was based on the comparison of cumulative upper respiratory tract symptoms scores (CURTS) in the asthmatic subjects treated with omalizumab compared to those treated with placebo over the first 4 days of acute infection. The symptoms evaluated daily included runny nose, sneezing, nasal congestion, sore throat, headache, chills/fever, fatigue, itchy/watery eyes. Symptom scores were recorded by subjects twice daily (in the morning and evening). Each symptom was scored on a scale of 1 to 3. Therefore, the total maximum (worst) score for a day would be 48. The scores recorded daily could range from 0 to 48.
Time Frame: 4 days
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mild Asthmatics Treated With Omalizumab | Mild Asthmatics Treated With Placebo Medication
Number analyzed (Participants) | 10 | 10
units on a scale | 20.2 [7.2 to 33.2] | 27.9 [17.1 to 38.7]
Statistical Analysis 1: Comparison: Mild Asthmatics Treated With Omalizumab vs Mild Asthmatics Treated With Placebo Medication; Test type: Superiority; p = 0.6, 2-sample t-test with unequal variances

6. Secondary Outcome: Number of Participants Whose FEV1 Dropped by More Than 20% During the Infection.
Description: Number of participants whose FEV1 dropped by more than 20% during the infection compared to their FEV1 value at baseline at the time of enrollment.
Time Frame: 21 days
Population: Two participants in the omalizumab treatment arm had to be dropped according to protocol because 1 developed a positive qPCR test for rhinovirus 4 weeks before virus inoculation, and the other developed a positive qPCR test for rhinovirus during the week before inoculation.
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Asthmatics Treated With Omalizumab | Mild Asthmatics Treated With Placebo Medication
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

7. Post Hoc Outcome: Time to Peak Airway Symptoms (Lower Respiratory Tract) Following Virus Inoculation.
Description: Time to peak airway symptoms (lower respiratory tract) following virus inoculation was compared among the asthmatics in the omalizumab treatment arm compared to time to peak symptoms among those in the placebo treatment arm.
Time Frame: 21 days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: days
Arm/Group | Mild Asthmatics Treated With Omalizumab | Mild Asthmatics Treated With Placebo Medication
Number analyzed (Participants) | 10 | 10
days | 16.0 [12.74 to 20.09] | 7.77 [4.61 to 13.07]
Statistical Analysis 1: Comparison: Mild Asthmatics Treated With Omalizumab vs Mild Asthmatics Treated With Placebo Medication; Test type: Superiority; p = 0.037, 2-sample t-test on the log scale — The p value is based on the fold change (ratio) of the geometric means of the time (days) to peak symptoms among asthmatics in the omalizumab/placebo treatment groups

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Mild Asthmatics Treated With Omalizumab | Mild Asthmatics Treated With Placebo Medication
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 5/15 | 4/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Asthmatics Treated With Omalizumab (N=15) | Mild Asthmatics Treated With Placebo Medication (N=16)
allergic rhinitis with hoarse voice (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Transient
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Transient
Anemia (low hemoglobin) (Blood and lymphatic system disorders) | 1 (1) | 2 (2) — Three subjects were dropped before the rhinovirus challenge. Their anemia was mild, but Hb level was < 10.0 gm/dL. They were seen by a doctor at the University of Virginia (student health).
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Transient
Insomnia (General disorders) | 1 (3) | 0 (0) — Episodic (3 times), but transient
Mild concusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Occurred during the Run-in period. Event causing the concussion was unrelated to the study.
Blood neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) — Blood neutropenia (< 1500 cells/mm3) occurred twice after rhinovirus was administered. The neutropenia resolved before the subject completed the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT02388997/Prot_SAP_000.pdf